CLINICAL TRIAL: NCT05456022
Title: Therapeutic Efficacy of Quercetin Versus Its Encapsulated Nanoparticle on Tongue Squamous Cell Carcinoma Cell Line
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hana'a Hezam Ghaleb Algadi, Ph.D. candidate at Oral &Maxillofacial Pathology Department- Faculty of Dentistry, Cairo University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 172022
Record Dates: First submitted 2022-06-25; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Oral Cancer
Keywords: Tongue; SCC; chemotherapy; Quercetin; PLGA-PEG nanoparticle
MeSH Terms: conditions — Mouth Neoplasms | interventions — Flavonoids; Quercetin; 4,6-dinitro-o-cresol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quercetin drug. (Experimental)
  Interventions: Drug: Quercetin 3,3',4',5,6-Pentahydroxyflavone, 2-(3,4-Dihydroxyphenyl)-3,5,7-trihydroxy-4H-1-benzopyran-4-one
- Quercetin-encapsulated PLGA-PEG nanoparticles (Experimental)
  Interventions: Drug: Quercetin-encapsulated PLGA-PEG nanoparticles (Nano-QUT)
- Doxorubicin chemotherapeutic drug (Active Comparator)
  Interventions: Drug: Doxorubicin chemotherapeutic drug as a positive control

INTERVENTIONS:
Drug: Quercetin 3,3',4',5,6-Pentahydroxyflavone, 2-(3,4-Dihydroxyphenyl)-3,5,7-trihydroxy-4H-1-benzopyran-4-one — Appearance (Color) Conforms Yellow Appearance (Form) Powder
  1H NMR Spectrum Conforms to Structure Loss on Drying < 4 % _ Purity (HPLC) > 95 %
  Other Names: Citrus bioflavonoid, Sophoretin; Meletin; Quercetine; Xanthaurine; Quercetol; Quercitin; Quertine; Flavin
  Arms: Quercetin drug.
Drug: Quercetin-encapsulated PLGA-PEG nanoparticles (Nano-QUT) — Nano QUT will prepared by PLGA-PEG nanocomposites that will be prepared by an oil-in-water (O/W) single emulsion solvent evaporation method
  Arms: Quercetin-encapsulated PLGA-PEG nanoparticles
Drug: Doxorubicin chemotherapeutic drug as a positive control — Doxorubicin is a type of chemotherapy drug called an anthracycline. It slows or stops the growth of cancer cells by blocking an enzyme called topo isomerase 2
  Arms: Doxorubicin chemotherapeutic drug

SUMMARY:
Squamous cell carcinoma (SCC) is the most common oral cavity carcinoma. Conventional therapeutic modalities for oral malignancy include surgery, radiotherapy and chemotherapy alone or in combinations.The major obstacle of using current anticancer drugs is; first the non-specific tissue distribution, as these drugs are unable to distinguish between normal and cancer cells.Quercetin is a bioactive flavonoid having strong antioxidant properties. .Among all the nanomaterials, polymeric nanoparticles are of significant interest for drug delivery applications due to many unique features of nanoparticle polymers.This is the first study to investigate the anticancer effects of (Quercetin) either free or encapsulated by PLGA-PEG NPs in tongue squamous cell carcinoma (TSCC) cell line.

DETAILED DESCRIPTION:
Squamous cell carcinoma (SCC) is the most common oral cavity carcinoma. Conventional therapeutic modalities for oral malignancy include surgery, radiotherapy and chemotherapy alone or in combinations. The major obstacle of using current anticancer drugs is; first the non-specific tissue distribution, as these drugs are unable to distinguish between normal and cancer cells. Quercetin is a bioactive flavonoid having strong antioxidant properties. It is naturally present in a wide variety of fruits and vegetables. Among all the nanomaterials, polymeric nanoparticles are of significant interest for drug delivery applications due to many unique features of nanoparticle polymers. Polymeric nanocarriers have been fabricated from natural and synthetic polymers. Poly ethylene glycol-poly lactide-co-glycolic acid (PEG-PLGA) amphiphilic copolymer is an emergent system because it can be easily synthesized and possesses a lot of good qualities. Several previous in vitro and in vivo studies have evaluated the cytotoxic effects of quercetin and have revealed that it decreases cell viability and increases cell apoptotic rate in OSCC. However, the anti-cancer property of quercetin in tongue squamous cell carcinoma (TSCC) has not been studied yet. This is the first study to investigate the anticancer effects of (Quercetin) either free or encapsulated by PLGA-PEG NPs in tongue squamous cell carcinoma (TSCC) cell line.

ELIGIBILITY:
Inclusion Criteria:

* Tongue Squamous cell carcinoma cell lines
* Quercetin drug.
* Quercetin-encapsulated PLGA-PEG nanoparticles (Nano-QUT)
* Application of a Quercetin drug as chemotherapeutic drug.
* Detection of Quercetin activity in apoptosis or cytotoxicity/cell viability.

Exclusion Criteria:

* Any cancer cell line other than tongue Squamous cell carcinoma cell lines
* Any use of Quercetin other than chemotherapy.
* Detection of Quercetin activities other than apoptosis or cytotoxicity/cell viability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000000 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cytotoxicity/Cell viability. | within 1 week after cell line propagation
  MTT assay for cellular viability:
  The cytotoxic impacts of the tested drugs and Nano QUT-encapsulation will be measured by MTT. The (HNO-97) cells will be cultured in 96-well plates at a density of 5 × 103 cells/well. All drugs with their described concentrations will be added to the media over tongue SCC cell lines. After a day of incubation, the dissolved MTT in PBS will be added to each well at a final concentration of 5 mg/ml, and the samples will be incubated at 37 °C for 4h. Water-insoluble dark blue formazan crystals that will be formed during MTT cleavage in actively metabolizing cells will then be dissolved in dimethyl sulfoxide (DMSO). Absorbance will be measured at A455 nm, using an ELISA microplate reader
Apoptosis. | within 1 week after cell line propagation
  Annexin V and propidium iodide (PI) stains will be used in the determination of apoptosis after treatment with the free, nano counterpart of QUT and free Dox post 24h of their incubation over the HNO-97 cell line. The apoptotic analysis will be dedicated to differentiating between early and late apoptotic cells, as well as necrotic cells. The apoptosis of the treated and untreated HNO-97 line with the proposed free, nano counterpart of Nano-QUT and Dox will be analyzed by ﬂow cytometer apparatus

SECONDARY OUTCOMES:
Gene expression of (BCL-2) . | within 1 week after cell line propagation
  Following treatment with the proposed free DOX, free and Nano-QUT formulations for 24 h, the cells are harvested, lysed and tested with RT-PCR using specific primers to estimate the fold change of the apoptotic signals (BCL-2 and Bax) and survival pathway (Expression of PI3K gene). GAPDH will be used as a housekeeping gene to normalize the level of target gene expression.
Gene expression of ( Bax gene) | within 1 week after cell line propagation
  Following treatment with the proposed free DOX, free and Nano-QUT formulations for 24 h, the cells are harvested, lysed and tested with RT-PCR using specific primers to estimate the fold change of the apoptotic Bax gene
survival pathway (Expression of pi3k gene) | within 1 week after cell line propagation
  Following treatment with the proposed free DOX, free and Nano-QUT formulations for 24 h, the cells are harvested, lysed and tested with RT-PCR using specific primers to estimate the fold change of survival pathway (Expression of pi3k gene)

CONTACTS AND LOCATIONS:
Locations (1):
- 11 Saraya El Manial, Cairo, Egypt